CLINICAL TRIAL: NCT00570635
Title: A Phase 2 Study of XL820 in Subjects With Advanced Gastrointestinal Stromal Tumors Resistant to or Intolerant of Imatinib and/or Sunitinib
Brief Title: A Phase 2 Study of XL820 in Adults With Advanced GIST Resistant to Imatinib and/or Sunitinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XL820-201
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-05

CONDITIONS: Gastrointestinal Stromal Tumors; Gastrointestinal Neoplasms
Keywords: GIST; Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: XL820
- B (Experimental)
  Interventions: Drug: XL820

INTERVENTIONS:
Drug: XL820 — XL820 capsules administered orally as a single agent at a dose of 800 mg daily
  Arms: A
Drug: XL820 — XL820 capsules administered orally as a single agent at a dose of 300 mg twice daily
  Arms: B

SUMMARY:
The purpose of this study is to evaluate the clinical benefit of the KIT inhibitor XL820 in subjects with advanced gastrointestinal stromal tumors (GIST) who are resistant to or intolerant of Imatinib and/or Sunitinib.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or locally advanced or unresectable GIST who have intolerance of or disease progression following prior treatment with imatinib and/or sunitinib
* ECOG (Eastern Cooperative Oncology Group) performance status ≤2
* Must have measurable disease per RECIST (Response Evaluation Criteria in Solid Tumors)
* Recovery from toxicity from prior therapy to Common Terminology Criteria for Adverse Events (CTCAE) v3.0 Grade ≤1 or to subject's baseline status
* Adequate organ and marrow function
* Sexually active subjects (male and female) must agree to use accepted methods of contraception during the course of the study and for 3 months following discontinuation of study drugs.
* Female subjects of childbearing potential must have a negative pregnancy test at enrollment.

Exclusion Criteria:

* Therapy with imatinib or sunitinib within 14 days before the first dose of study drug
* Chemotherapy, immunotherapy, targeted therapy, chemoembolization, or any investigational drug for the treatment of GIST after the last dose of imatinib or sunitinib
* Anticoagulation with warfarin or coumarin-related compounds
* Radiation to ≥25% of bone marrow within 28 days of study entry
* Treatment with other investigational agents within 28 days of the first dose of XL820
* Known central nervous systems metastases
* Uncontrolled or intercurrent illness
* Pregnancy or breast-feeding
* Active bacterial or viral infection requiring systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Clinical benefit, defined as either confirmed complete response, confirmed partial response, or evidence of stable disease lasting ≥16 weeks, in subjects with advanced GIST resistant to/intolerant of imatinib and/or sunitinib | Assessed at baseline, Week 4 and 8, and every 8 weeks thereafter

SECONDARY OUTCOMES:
Safety and tolerability of XL820 | Assessed at each visit
Progression-free survival, duration of response, and overall survival | Assessed until progression
Further characterize the pharmacokinetic and pharmacodynamic parameters of XL820 in subjects with advanced GIST | Assessed during periodic visits

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Los Angeles, California
  - Park Ridge, Illinois
  - Boston, Massachusetts